CLINICAL TRIAL: NCT02369731
Title: Long-Term Observational Study of Translarna Safety and Effectiveness in Usual Care
Brief Title: Registry of Translarna (Ataluren) in Nonsense Mutation Duchenne Muscular Dystrophy (nmDMD)
Status: Active, not recruiting | Type: Observational
Sponsor: PTC Therapeutics (Industry)
Collaborators: The John Walton Muscular Dystrophy Research Centre (TREAT-NMD) (Unknown); Cooperative International Neuromuscular Research Group (Network)
Responsible Party: Sponsor
Other Study IDs: PTC124-GD-025o-DMD
Record Dates: First submitted 2015-01-28; First posted 2015-02-24 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Translarna: Participants with nmDMD receiving Translarna will be followed for at least 5 years from their date of enrollment, or until participant withdrawal of consent or death, whichever occurs first.

SUMMARY:
This study is being performed as a post-approval safety study (PASS), per the Pharmacovigilance Risk Assessment Committee (PRAC) of the European Medicines Agency (EMA), to gather data on Translarna (ataluren) safety, effectiveness, and prescription patterns in routine clinical practice.

DETAILED DESCRIPTION:
This is a multicenter, observational study of participants receiving Translarna based on inclusion of their data in a registry. This study is intended to enroll 360 participants across ~50 care centers in Europe and other regions over a period of ~ 2 years. The study population will include participants who are receiving usual care treatment with commercial supply of Translarna (or receiving care within a named participant early access program) and who provide consent. Participants will be followed for at least 5 years from their date of enrollment. Safety and efficacy data will be collected in conjunction with routine visits conducted as per usual care. Although there are no protocol-mandated procedures, it is expected that physicians and other caregivers will follow published treatment guidelines and standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Receiving or will be receiving usual care treatment with commercial supply of Translarna (or receiving care within a named participant early access program)
* Willing to provide written informed consent to allow the study data collection procedures (either by the participant or through authorisation by a legal guardian)

Exclusion Criteria:

* Participants who are receiving ataluren or placebo in a blinded, randomized clinical trial, or ataluren in any other ataluren clinical trial or cohort early access program that prevents participation in this study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target study population will include participants for whom the decision to prescribe Translarna (outside of a clinical trial) has already been made, including participants in named participant early access programs. Participants within each prescriber's practice who are or will be receiving treatment with Translarna, and who meet the eligibility criteria and provide informed consent (either by the participant or through authorisation by a legal guardian) will be invited to enroll into the study and will be followed according to the protocol.
Sampling Method: Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | 5 years

SECONDARY OUTCOMES:
Prescriber and Participant Compliance With Prescribing Information According to the Approved Labelling | 5 years

OTHER OUTCOMES:
Participant Health Management Measures | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Johnson, Study Director — PTC Therapeutics
Locations (71):
- Austria (2):
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - Sozialmedizinisches Zentrum Süd Kaiser-Franz-Josef Spital mit Gottfried von Preyer´schen Kinderspital, Vienna
- Hospital das Clínicas da Universidade de São Paulo, São Paulo, Brazil
- Czechia (2):
  - The University Hospital Brno, Brno
  - Motol University Hospital, Praha 5 - Motol
- France (17):
  - CHU de Bordeaux Hôpital Pellegrin Enfant, Bordeaux
  - CHRU de Brest Hôpital Morvan, Brest
  - Hospices Civils de Lyon Groupement Hospitalier Est - Bâtiment "Les Tilleuls", Bron
  - CHU de Clermont-Ferrand, hôpital Estaing, Clermont-Ferrand
  - CHU de Martinique - Hôpital P. Zobda-Quitman, Fort de France Cedex
  - CHRU de Lille, Lille
  - CHU de Marseille Hôpital de la Timone, Marseille
  - CHU de Nantes, Nantes
  - Hôpital Armand Trousseau, Paris
  - Hôpital Necker - Enfants malades, Paris
  - CHU de Reims American Memorial Hospital, Reims
  - CHU de Saint-Etienne Hôpital Bellevue, Saint-Etienne
  - CHU de la Réunion - GHSR - GH Sud-Réunion, Saint-Pierre
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse Hôpital Pierre Paul Riquet, Toulouse
  - CHRU de Tours Hôpital Bretonneau, Tours
  - CHU de Nancy Hôpital de Brabois-Enfants Rue du Morvan, Vandœuvre-lès-Nancy
- Germany (10):
  - Klinikum Bayreuth GmbH, Bayreuth
  - Sozialpädiatrisches Zentrum (SPZ) Charité Berlin, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Essen (AoR), Essen
  - SPZ Frankfurt Mitte, Frankfurt am Main
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - MVZ Kinder- und Jugendärzte Fürth GmbH, Fürth
  - Universitätskinderklinik Gießen, Giessen
  - Klinik und Poliklinik f. Kinder- und Jugendmedizin, Hamburg
  - Muskelzentrum, Schwerpunkt Neuropädiatrie, Kassel
- Greece (2):
  - Children's Hospital "Aghia Sophia", Athens
  - Ahepa University Hospital, Thessaloniki
- Hungary (2):
  - Semmelweis Egyetem II (Semmelweis University II), Budapest
  - Szent László Kórház Gyermekneurológiai szakrendelés, Budapest
- Israel (3):
  - Hadassah Mount Scopus Medical Center, Jerusalem
  - Schneider Medical Center Tel Aviv University, Petah Tikva
  - Sheba Medical Center The Joseph Sagol EMG, Neuroscience Center, Ramat Gan
- Italy (12):
  - IRCSS Istituto delle Scienze Neurologiche, Bologna
  - Istituto Giannina Gaslini, Genova
  - AOU Policlinico "G. Martino", Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Istituto Neurologico Carlo Besta, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - II Policlinico Neurofisiopatologia (Edificio 11 G), Napoli
  - Cardiomiologia e Genetica Medica Primo Policlinico, Napoli
  - AO Padova Clinica Neurologica, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Bambino Gesù Children's Hospital, Rome
  - Ospedale Molinette SCDU Neuropsichiatria Infantile AO Città della Salute e della Scienza di Torino, Torino
- Bērnu klīniskā universitātes slimnīca, Riga, Latvia
- St. Olavs hospital University children's clinical hospital, Trondheim, Norway
- Portugal (3):
  - Centro Hospitalar e Universitário de coimbra EPE - Hospital Pediátrico de Coimbra, Coimbra
  - Centro Hospitalar Lisboa Norte EPE - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto EPE - Hospital Geral de Santo António, Porto
- Romania (2):
  - Spitalul Clinic de Copii "Dr. Victor Gomoiu" Sectia Clinica Neurologie Pediatrica, Bucharest
  - Regina Maria Policlinica Opera Center, Bucharest
- University Children's Hospital University Medical Centre Ljubljana, Ljubljana, Slovenia
- Sweden (2):
  - Göteborgs Universitet Avdelningen för pediatrik vid institutionen för kliniska vetenskaper, Gothenburg
  - Karolinska Institutet, Stockholm
- United Kingdom (10):
  - Birmingham Heartlands Hospital, Birmingham
  - Bristol Children's Hospital, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Children Hospital - Children's Neurosciences Leeds TEACHING HOSPITALS NHS Trust, Leeds
  - Children's Hospital Alder Hey Children's Hospital NHS Trust, Liverpool
  - St Thomas' Hospital Children Services, London
  - UCL Great Ormond Street Institute of Child Health, London
  - Royal Manchester Children's Hospital, Manchester
  - The John Walton Muscular Dystrophy Research Centre, Newcastle
  - NIHR Lancashire Clinical Research Facility Royal Preston Hospital, Preston

REFERENCES:
- [Derived] Mercuri E, Osorio AN, Muntoni F, Buccella F, Desguerre I, Kirschner J, Tulinius M, de Resende MBD, Morgenroth LP, Gordish-Dressman H, Johnson S, Kristensen A, Werner C, Trifillis P, Henricson EK, McDonald CM; STRIDE and CINRG DNHS investigators. Safety and effectiveness of ataluren in patients with nonsense mutation DMD in the STRIDE Registry compared with the CINRG Duchenne Natural History Study (2015-2022): 2022 interim analysis. J Neurol. 2023 Aug;270(8):3896-3913. doi: 10.1007/s00415-023-11687-1. Epub 2023 Apr 28. PMID 37115359
- [Derived] Mercuri E, Muntoni F, Osorio AN, Tulinius M, Buccella F, Morgenroth LP, Gordish-Dressman H, Jiang J, Trifillis P, Zhu J, Kristensen A, Santos CL, Henricson EK, McDonald CM, Desguerre I; STRIDE; CINRG Duchenne Natural History Investigators. Safety and effectiveness of ataluren: comparison of results from the STRIDE Registry and CINRG DMD Natural History Study. J Comp Eff Res. 2020 Apr;9(5):341-360. doi: 10.2217/cer-2019-0171. Epub 2020 Jan 30. PMID 31997646